CLINICAL TRIAL: NCT02667522
Title: Targeting Biomarkers of Risk for Depression and Anxiety Through a Parenting Intervention
Brief Title: Shaping Neural Activity Through Parenting
Acronym: SNAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Kristin Bernard, Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21MH108766-01A1 (NIH)
Record Dates: First submitted 2016-01-11; First posted 2016-01-29 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parenting Intervention (Experimental): Parenting Intervention: Parent-Child Interaction Therapy (PCIT)
  Interventions: Behavioral: Parent Child Interaction Therapy (PCIT)
- Waitlist Control (No Intervention): Waitlist Control Condition

INTERVENTIONS:
Behavioral: Parent Child Interaction Therapy (PCIT) — PCIT includes 12-16 sessions across two phases: the first focused on enhancing positive parenting during child-directed interactions, and the second focused on reducing harsh parenting during parent-directed interactions. Parents receive feedback and coaching on their interactions with the child during sessions.
  Arms: Parenting Intervention

SUMMARY:
The purpose of this study is to test causal links between dimensions of positive and harsh parenting and children's brain responses to rewards and errors, using a parenting intervention.

DETAILED DESCRIPTION:
Depression and anxiety are among the most frequently diagnosed psychological disorders, with persistent patterns of impairment evident from childhood through adulthood. Impaired functioning of core brain systems that respond to reward and errors may increase risk for depression and anxiety. Importantly, these neural risk markers for depression and anxiety appear to be shaped, at least in part, by environmental input. Problematic parenting is a key environmental factor involved in the intergenerational transmission of depression and anxiety. Low positive parenting is associated with blunted brain responses to reward and harsh parenting is associated with heightened brain responses to errors. This study uses an evidence-based parenting program to test causal links between dimensions of positive and harsh parenting and children's brain responses to rewards and errors. Participants will include 80 6- to 7-year-old children and their mothers who will be randomly assigned to participate in a parenting program (Parent Child Interaction Therapy: PCIT) or to a waitlist control group, and brain responses to rewards and errors will be assessed pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Child is 6-7 years old
* Maternal history of anxiety or depression
* Maternal self-report of low positive/high harsh parenting

Exclusion Criteria:

* Child has developmental disorder

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Event-Related Potentials (ERP) | On average, 1 month after intervention
  ERP responses to reward (i.e., feedback negativity) and errors (i.e., error-related negativity)

SECONDARY OUTCOMES:
Parenting quality | On average, 1 month after intervention
  Observational assessments of positive and harsh parenting
Child anxiety symptoms | On average, 1 month after intervention
  Parent Questionnaire
Child depressive symptoms | On average, 1 month after intervention
  Parent Questionnaire
Child anxiety | On average, 1 month after intervention
  Structured diagnostic interview
Child depression | On average, 1 month after intervention
  Structured diagnostic interview

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Bernard, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided